CLINICAL TRIAL: NCT06674499
Title: A Randomized Controlled Clinical Trial on the Development and Evaluation of a Self-Management Model for Cancer Rehabilitation
Brief Title: Development and Evaluation of a Self-Management Model for Cancer Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xingchen Peng (Other)
Responsible Party: Sponsor-Investigator, Xingchen Peng, Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-1567
Record Dates: First submitted 2024-10-28; First posted 2024-11-05 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Cancer; Rehabilitation; Psychotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-help rehabilitation model (Experimental)
  Interventions: Other: Self-help rehabilitation model
- Conventional rehabilitation model (Placebo Comparator)
  Interventions: Other: Conventional rehabilitation model

INTERVENTIONS:
Other: Self-help rehabilitation model — The intervention measures followed the principles and processes of cognitive-behavioral therapy. Three intervention sessions were conducted over a period of eight weeks. The first session lasted 90 minutes, while the subsequent sessions (in weeks 4 and 8) lasted 45 minutes each and were conducted face-to-face by the therapist.
  Arms: Self-help rehabilitation model
Other: Conventional rehabilitation model — The control group, which follows the conventional rehabilitation model, operates under the current standard of cancer treatment and follow-up. In this model, oncology healthcare professionals provide recommendations based on the specific circumstances of the patients. However, the choice of the rehabilitation model is primarily decided by the patients themselves, aligning with current clinical practice.
  Arms: Conventional rehabilitation model

SUMMARY:
Participants were primarily recruited from medical institutions, specifically targeting newly diagnosed patients with malignant tumors. They were randomly assigned to two different rehabilitation models using block randomization: the cancer self-help rehabilitation model or the conventional rehabilitation model.

During the intervention period, trained oncology advanced practice nurses conducted weekly questionnaire surveys for enrolled patients. During the follow-up period, these surveys were conducted every four weeks. Peripheral venous blood samples were collected at baseline and at weeks 0, 4, 8, and 12 after the intervention began to test for biomarkers related to emotional distress.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed with head and neck malignancy.
* Experiencing psychological distress.
* Aged between 18 and 70 years.
* Patients scheduled to receive antitumor treatment in a day hospital or outpatient setting.
* ECOG performance status score of 0-2.
* Patients voluntarily participate, fully understand, and are able to independently complete the questionnaires.

Exclusion Criteria:

* A history of other malignancies within the past 5 years.
* A history of any mental illness, including but not limited to: generalized anxiety disorder, depressive disorder, panic disorder, schizophrenia, or bipolar disorder.
* Patients currently receiving other psychological treatments or taking psychiatric medications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Degree of improvement in emotional distress | 16 weeks
  After the intervention period for the patients, the change in the HADS (Hospital Anxiety and Depression Scale) total score was assessed based on the scoring criteria, comparing the scores to the baseline.
  The HADS scoring ranges are as follows:
  Total Score Range: 0 to 42； Anxiety Subscale (HADS-A): 0 to 21； Depression Subscale (HADS-D): 0 to 21；
  Score Interpretation:
  0-7: Normal range, typically indicating no significant anxiety or depression symptoms.； 8-10: Mild anxiety or depression, may warrant monitoring; 11-14: Moderate anxiety or depression, further assessment or intervention is advisable; 15 and above: Severe anxiety or depression, usually requiring professional mental health intervention; In summary, higher scores on the HADS indicate more severe symptoms of anxiety or depression.

SECONDARY OUTCOMES:
Levels of improvement in quality of life | 16 weeks
  The QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30) is a tool designed to assess the quality of life in cancer patients. It consists of 30 items covering various dimensions of quality of life, including functional status, symptoms, and overall health status.
  Score Range:
  Functional Status:
  Maximum Score: 100 Minimum Score: 0.
  Symptoms:
  Maximum Score: 100 (note: higher scores indicate worse symptoms) Minimum Score: 0.
  Overall Health Status:
  Maximum Score: 100 Minimum Score: 0.
  Evaluating Treatment Effects: Comparing scores before and after treatment to assess the impact on quality of life.
  Clinical Research: As a standard tool for assessing quality of life in cancer studies.
  Patient Management: Helping healthcare providers identify specific patient needs to optimize treatment plans.
Levels of anxiety and depression | 16 weeks
  Anxiety and Depression: Assessed at baseline (before intervention), every two weeks during the intervention period, and every four weeks during the follow-up period, according to the scoring criteria of the HADS.
  Score Range Maximum Score: Each subscale has a maximum score of 21 (7 items × 3 points each).
  Minimum Score: Each subscale has a minimum score of 0 (indicating no symptoms).
Levels of Supportive care needs | 16 weeks
  Supportive Care Needs Level: Evaluated at baseline (before intervention), every two weeks during the intervention period, and every four weeks during the follow-up period, using the scoring criteria of the Supportive Care Needs Survey (SCNS-SF34).
  Scoring Method: Each item is typically rated on a 4-point Likert scale (1 = no need, 2 = low need, 3 = moderate need, 4 = high need).
  Total Score Range:Minimum Score: 34 (if every item is scored as 1)；Maximum Score: 136 (if every item is scored as 4)。 Score Significance 34-68: Low Need; Indicates that the patient has minimal supportive care needs. 69-102: Moderate Need; Suggests that the patient has some areas where additional support or resources may be beneficial.
  103-136: High Need; Reflects significant supportive care needs across multiple domains, indicating that the patient may require urgent intervention and comprehensive support.

OTHER OUTCOMES:
Levels of Peripheral stress biomarkers | 16 weeks
  Peripheral venous blood samples were collected from enrolled patients at baseline and at weeks 0, 4, 8, and 12 after intervention. The stress biomarkers tested include the concentrations of adrenaline, norepinephrine, cortisol, and adrenocorticotropic hormone. The patient needs to lie on their back for 15 minutes before blood collection, and must avoid drinking alcohol, coffee, and smoking for 12 hours before blood collection. After collection, the blood sample should be immediately sent to the laboratory for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- WestChina Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No